CLINICAL TRIAL: NCT06484543
Title: Brown Fat as Therapeutic Strategy for Obesity and Associated Metabolic Diseases Via Functional/Nutraceutical Approach - Molecular Mechanisms of Pentacyclic Triterpenes (BRACE)
Brief Title: Brown Fat as Therapeutic Strategy for Obesity and Associated Metabolic Diseases Via Functional Food/Nutraceutical Approach - Molecular Mechanisms of Pentacyclic Triterpenes (BRACE)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Human Development and Potential (IHDP), Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Principal Investigator, Melvin Leow, Principal Investigator, Institute for Human Development and Potential (IHDP), Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2024/00022
Record Dates: First submitted 2024-06-04; First posted 2024-07-03 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Diabetes; Brown Adipose Tissue
MeSH Terms: conditions — Diabetes Mellitus | interventions — maslinic acid

STUDY DESIGN:
Intervention Model Description: Single blinded study
Who Masked: Participant
Masking Description: This is a single-blind study in which the participants will not know which group will be assigned to and only the investigators will know.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maslinic Acid (Experimental): MA (an extract from olive fruit). Each participant will be instructed to take 3 tablets (60 mg or equivalent) daily after breakfast for 12 weeks.
  Interventions: Other: Maslinic Acid
- Placebo (Placebo Comparator): Each subject will be instructed to take 3 matching placebo tablets (or equivalent) daily after breakfast for 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Maslinic Acid — Consumption of Maslinic Acid for 12 weeks
  Arms: Maslinic Acid
Other: Placebo — Consumption of Placebo for 12 weeks
  Arms: Placebo

SUMMARY:
To examine MA (Maslinic Acid) safety and efficacy in ameliorating insulin resistance and the cardinal features of metabolic syndrome. Chronic exposure to MA as a potent PPARgamma binder nutraceutical over 12 weeks will result in improvement in the features of metabolic syndrome including waist circumference, blood pressure, serum HDL-C level, fasting serum triglycerides and fasting plasma glucose. Expected secondary endpoints include favorable changes in metabolic rate, respiratory quotient, fat oxidation, body composition, weight, BAT/WAT compartments, batokines/adipokines, proinflammatory biomarkers, insulin sensitivity and beta cell function.

DETAILED DESCRIPTION:
Up to 50 participants that are overweight/obese people suffering from metabolic syndrome/pre-metabolic syndrome will be recruited for this study. They will be asked to come to the Clinical Nutrition Research Centre (CNRC) for a screening session (1st visit) and given plenty of time to read this information sheet and the opportunity to ask questions. Once they are fully informed regarding the study and all their questions have been satisfactorily answered, they will be given a consent form to complete and sign in the presence of the researcher. Following this, in order to gauge their suitability for taking part in the study, an assessment will be carried out. This assessment needs to be carried out in a fasted state and they would therefore have to come one morning following an overnight fast. The screening will include anthropometric measurements, blood pressure measurement and blood sampling. Anthropometric measurements taken will be height, weight, waist circumference and hip circumference. Body composition will be measured using an electrical impedance analyser (BIA). Blood pressure will be measured using an automatic blood pressure monitor. They will also undergo a blood sampling from their vein (6 mL or approximately 1.5 teaspoons) to be tested for thyroid function, glucose and lipid profile. Once they have been accepted into the study, they will then be expected to come to the centre for a total of four separate test sessions, over a span of approximately 3 months (two test sessions each at week 0 (before intervention) and at week 12 (after intervention) which will be scheduled within 4 weeks from each timepoint) and will be randomly assigned (via www.random.org) to either the MA or placebo groups below (up to 25 subjects per group). This is a single-blind study in which the participants will not know which group will be assigned to and only the investigators will know. After completing the two test sessions for week 0, both groups will start consuming either the 60mg of MA or placebo once (depending on which group they are assigned to) daily after breakfast for 12 weeks. For each of the four test sessions, they will be required to fast overnight and avoid caffeine and alcohol for 8-10 hours before reporting at the CNRC in the morning between 8 to 9 AM. Only plain water can be consumed during the fast. They are to avoid any physical activity/exercise and alcohol on the day prior to the visit. The test sessions will be as follows: On the first test session (2nd visit) at week 0 (before intervention), they will need to come to CNRC in the morning in a fasted state and an intravenous indwelling cannula will be inserted into an arm vein to collect a fasting blood sample (40ml or approximately 8 teaspoons) and an urine sample will also collected. They will then proceed to undergo metabolic rate measurement with IRT focusing on their neck and area above the collar bone in a whole body room calorimeter (WBC) for the next 45 minutes. They will then undergo a mild cold stimulation of about 14 degree Celcius by wearing a cooling vest for the next 1.5 hours, in which metabolic rate measurement and IRT in the WBC will be performed during this period. Wearing the cooling vest may lead to some shivering, but it is generally considered safe. Upon exiting the WBC, they will remove the cooling vest and 20ml (approximately 4 teaspoons) of blood sample and another urine sample will be collected again. After which, they will be free to leave.On the second test session (3rd visit) at week 0 (before intervention), they will need to come to CNRC in the morning in a fasted state and anthropometric measurements like height, weight, waist circumference and hip circumference will be taken. Body composition will be measured using an electrical impedance analyser (BIA) and blood pressure will be measured using an automatic blood pressure monitor. They will then undergo a body composition evaluation using dual energy X-ray absorptiometry (DXA) (approximately 20 mins duration) which allows quantification of fat, lean and bone mass. After that, an intravenous indwelling cannula will be inserted into an arm vein to collect a fasting (timepoint 0min) blood sample (5ml or approximately 1 teaspoon). Subsequently they will undergo a 120-minutes oral glucose tolerance test (OGTT) where you will be required to consume a glucose drink (75g of glucose) within 5 minutes. Following the consumption of the glucose drink, we will take further blood samples (from the cannula) every 30 minutes for the remaining 120 minutes (4 timepoints at 30, 60, 90 and 120 min). At each time point, approximately 5 ml or approximately 1 teaspoon of blood will be drawn.

During the entire test session, they will have to stay rested and in the laboratory. Television and a workspace will be provided for their use if they require. At the end of 2 hours of testing, they will be free to leave. The above 2 test sessions may be scheduled in any order, but to be completed no more than 4 weeks apart. They will now start the study intervention for the next 12 weeks. Depending on which group they are assigned to, they will be instructed to consume either 60mg of MA or placebo daily (after breakfast) for the next 12 weeks. They will then be required to come for the third test session (4th visit) and fourth test session (5th visit) at week 12 (after completing the 12 weeks of intervention), and repeat the same procedures as per that of the first test session (2nd visit) and the second test session (3rd visit) respectively. The 2 test sessions each at week 0 and 12 may be scheduled within 4 weeks from each time point. During the course of the study, there is a possibility that we might unintentionally come to know of new information about their health condition from (e.g. the screening blood test, etc.) that are conducted as part of the study. These are called "incidental findings". "Incidental findings" are findings that have potential health or reproductive importance to research participants like you and are discovered in the course of conducting the study, but are unrelated to the purposes, objectives or variables of the study. These findings may affect your current or future life and/or health insurance coverage. Examples of potential incidental findings that may be discovered during the course of this study may include but are not limited to greater than normal range of fasting glucose, insulin, C-peptide or HbA1C (possibly indicating type 2 diabetes), abnormal lipid profile (e.g., high triglycerides) or thyroid hormones (e.g. TSH, FT4). Incidental finding (IF) management workflow:- Participants will be asked during informed consent if they would like to be re-identified and re-contacted in the event of an incidental finding (IF) during the course of future research. Study participant wishes on the return of IF are documented in the informed consent form utilized by the study team. - A list of coded study IDs who have indicated their wish on the return of IF will be provided to the PI.- The PI will evaluate the findings with a competent and qualified clinician/healthcare professional/ study doctor. The PI will confirm against the consent form that the participant had indicated their wishes to be re-identified and re-contacted in the event of an IF. If so, the study participant will be de-identified by the PI to contact the participant.- The PI (or his/her study team) will re-contact the participant and re-confirm if participant would like to be informed of the IF. The IF and its relevant information will be provided to the participant according to their preferred manner (either electronically or physical copy). They will be advised to seek a medical practitioner for further evaluation to reconfirm the IF. In the event that the participant is non-contactable, the study team will need to demonstrate and document that reasonable efforts have been made to re-contact the participant or next of kin. The PI (or his/her study team) will document the above in the study records. The PI (or his/her study team) will also update study folder that the loop has been closed.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Chinese ethnicity
* Age between 21 to 60 years• Able to give informed consent
* Body mass index (BMI) between 23 to 32 kg/m2
* Thyroid function test must be within the normal ranges
* Willing to avail yourself for the whole study and follow study procedures
* EITHER deemed to have pre-metabolic syndrome when waist circumference is > 90 cm in men or > 80 cm in women, with none or up to one of the following condition:

  1. Triglyceride level >/= 1.7 mmol/L
  2. HDL cholesterol </= 1.0 mmol/L in men, and </= 1.3 mmol/L in women
  3. Blood pressure >/= 130/85 mmHg
  4. Fasting blood glucose >/= 6.1 mmol/L
* OR deemed to have metabolic syndrome when three or more of the following conditions are present:

  1. Waist circumference > 90 cm in men and > 80 cm in women
  2. Triglyceride level >/= 1.7 mmol/L
  3. HDL cholesterol</= 1.0 mmol/L in men, and </= 1.3 mmol/L in women
  4. Blood pressure >/= 130/85 mmHg
  5. Fasting blood glucose >/= 6.1 mmol/L

Exclusion Criteria:

* Are pregnant or contemplating pregnancy (for female subjects)
* Partake in sports at the competitive and/ or endurance levels
* Have known glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Have major chronic disease such as heart disease or cancer
* Take insulin or drugs known to affect glucose metabolism
* Intentionally restrict food intake
* Have major medical or surgical event requiring hospitalization within the preceding 3 months
* Have taken antibiotics for 3 months before the study period
* Are a smoker
* Are an overnight shift worker
* Have any known food allergy (eg. anaphylaxis to peanuts) or skin allergy (eg. rashes due to alcohol, etc)
* Having active Tuberculosis (TB) or currently receiving treatment for TB
* Have any known Chronic Infection or known to suffer from or have previously suffered from or is a carrier of Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), Human Immunodeficiency Virus (HIV)
* Are a member of the research team or their immediate family members. Immediate family member is defined as a spouse, parent, child, or sibling, whether biological or legally adopted
* Enrolled in a concurrent research study judged not to be scientifically or medically compatible with this study
* Have poor veins impeding venous access
* Have any history of severe vasovagal syncope (blackouts or near faints) following blood draws
* History of claustrophobia

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Concentration of blood glucose | Week 0, 12
Rate of brown adipose tissue activation detection using Infrared camera | Week 0, 12
Change in Energy Expenditure using Whole Body Calorimeter | Week 0, 12
Change in Body Mass Index (BMI) | Week 0, 12
  Measurement of weight and height
Change in Fat percentage | Week 0, 12
Concentration of Insulin level | Week 0, 12

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore Institute of Clinical Sciences, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No